CLINICAL TRIAL: NCT03019367
Title: Premature Infants Receiving Milking or Delayed Cord Clamping: Randomized Controlled Multicenter Non-inferiority Trial
Brief Title: Premature Infants Receiving Milking or Delayed Cord Clamping: PREMOD2
Acronym: PREMOD2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Collaborators: Sharp Mary Birch Hospital for Women & Newborns (Other); Loma Linda University (Other); University of Pittsburgh (Other); Providence Hospital (Other); University of Alabama at Birmingham (Other); University of Alberta (Other); University College Cork (Other); University of Ulm (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Christiana Care Health Services (Other); Sharp Grossmont Hospital (Other); University of Utah (Other); University of Mississippi Medical Center (Other); PIH Health Good Samaritan Hospital (Unknown); University of California, Irvine (Other); Children's Hospital Medical Center, Cincinnati (Other); Cook County Health (Other Government); St. Louis University (Other); LAC+USC Medical Center (Other)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director of Neonatal Research Institute, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PREMOD2; 1R01HD088646-01A1 (NIH)
Record Dates: First submitted 2016-11-21; First posted 2017-01-12 (Estimated); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Intraventricular Haemorrhage Neonatal; Death; Neonatal
Keywords: Premature infants; Umbilical cord milking; Delayed cord clamping; Intraventricular Hemorrhage; Death
MeSH Terms: conditions — Perinatal Death; Premature Birth; Death | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: It is not possible to blind the delivering obstetrician, however all other caregivers will be blinded. The procedure will be documented as "placental transfusion" in the delivery summary or admission-progress notes and all study assessments whether primary (head US) or secondary (neurodevelopmental exams) will be performed by blinded team members.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical cord milking UCM (Active Comparator): Milking the umbilical cord 4 times towards the infant at a speed of 20cm/2seconds.
  Interventions: Procedure: Umbilical cord milking UCM
- Delayed cord clamping DCC (Active Comparator): Delayed clamping of the umbilical cord for at least 60 seconds.
  Interventions: Procedure: Delayed cord clamping DCC

INTERVENTIONS:
Procedure: Umbilical cord milking UCM — At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before it is clamped. This procedure infuses a placental transfusion of blood into the preterm neonate and can be done in 15-20 seconds.
  Arms: Umbilical cord milking UCM
Procedure: Delayed cord clamping DCC — At delivery, delayed cord clamping will be performed by having the delivering obstetrician delay clamping of the umbilical cord for at least 60 seconds.
  Arms: Delayed cord clamping DCC

SUMMARY:
This study is being done to find out whether umbilical cord milking (UCM) is at least as good as or better than delayed cord clamping (DCC) to reduce bleeding in the brain or prevent death in premature newborns. The investigators will study short and long term outcomes of infants delivered before 32 weeks gestation that receive either UCM or DCC.

* The trial was stopped by the DSMB for safety in the small strata. They subsequently allowed for continuation of the trial in infants 29-32+6 wk GA.

DETAILED DESCRIPTION:
Aim 1. Compare the incidence of severe intraventricular hemorrhage (IVH) and/or death in premature newborns <33 weeks gestational age (GA) delivered by C/S receiving UCM to those receiving DCC.

Hypothesis1: First demonstrate infants in the UCM group are not inferior to the DCC group (reject H10).

Hypothesis2: If H1 is true, demonstrate lower incidence of severe IVH and/or death in UCM infants compared to DCC.

Aim 2. Compare the safety and efficacy profiles of premature newborns <33 weeks GA delivered by C/S receiving UCM vs. DCC during their hospitalization.

Hypothesis3: UCM group will have a decreased need for resuscitation interventions with no differences in bilirubin or polycythemia compared to DCC.

Hypothesis4: UCM group will have improved blood pressures in the first 24 hours of life compared to DCC.

Aim 3 (exploratory). To compare the outcomes of premature newborns <33 weeks GA delivered by C/S (Cesarean section) (from Aims 1 and 2) with those born by V/D (vaginal delivery) receiving UCM or DCC.

ELIGIBILITY:
Inclusion Criteria:

* 23 to 32 +6 Gestational age (currently enrolling 29 to 32+6 weeks)
* Multiples without Twin-to-twin Transfusion Syndrome (TTTS)

Exclusion Criteria:

* Congenital anomalies
* Major cardiac defects
* Placental abruption or previa with hemorrhage
* Cord prolapse
* Hydrops
* Bleeding Accreta
* Monochorionic multiples with evidence of TTTS
* Fetal or maternal risk (i.e. compromise)
* Parents declined study
* Unlikely to return for 2 yr Follow Up

Ages: 23 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1201 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Incidence of severe IVH or death | Through study completion at death or discharge, up to 6 months corrected gestational age (CGA)
  Severe intraventricular hemorrhage of grade 3 or 4 or death

SECONDARY OUTCOMES:
All Grade IVH | Through study completion at discharge, up to 6 months corrected gestational age (CGA)
  Any intraventricular hemorrhage (grades 1-4)
Severe IVH (Grade 3 or 4) | Through study completion at discharge, up to 6 months corrected gestational age (CGA)
  Severe intraventricular hemorrhage (bleeding in the brain parenchyma and/or ventricular dilation)
Hemoglobin/Hematocrit at 4 hours | 4 +/- 2 hours of life
  hemoglobin/hematocrit
Incidence of Severe IVH or death in infants <28 weeks gestation | Through study completion at discharge, up to 6 months corrected gestational age (CGA)
  Severe intraventricular hemorrhage (grade 3 or 4) in infants born under 28 weeks gestational age
Delivery room interventions | In the first 10 minutes of life
  Resuscitation interventions including positive pressure ventilation, continuous positive airway pressure, intubation, chest compressions and medications
Blood pressures in the first 24 hours of life | In the first 24 hours of life
  Blood pressure on admission, 6, 12, 18 and 24 hours of life

CONTACTS AND LOCATIONS:
Overall Officials: Anup C Katheria, MD, Principal Investigator — Sharp HealthCare
Locations (18):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - Loma Linda Medical Center, Loma Linda, California
  - LAC+USC Medical Center, Los Angeles, California
  - PIH Health Good Samaritan Hospital, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - Sharp Grossmont Hospital, San Diego, California
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California
  - Christiana Care, Newark, Delaware
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Louis University, St Louis, Missouri
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Governors of University of Alberta, Edmonton, Alberta, Canada
- University of ULM, Ulm, Baden-Wurttemberg, Germany
- Cork University Maternity Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available per NICHD requirements (National Institute of Child Health and Human Development).
Supporting Information: SAP
Time Frame: 2 years after primary publication
Access Criteria: An archived dataset with documentation will be made available for additional uses by outside investigators, in collaboration with the study investigators. We will work with NICHD program staff to develop a broad data sharing plan over time.

REFERENCES:
- [Derived] Katheria AC, Allman P, Szychowski JM, Essers J, Carlo WA, Schmolzer GM, Dempsey E, Yanowitz T, Kaempf J, Vora F, Bhat S, Arnell K, Rich W, Varner M. Perinatal Outcomes of Subjects Enrolled in a Multicenter Trial with a Waiver of Antenatal Consent. Am J Perinatol. 2022 Jun;39(8):904-908. doi: 10.1055/s-0040-1719184. Epub 2020 Nov 3. PMID 33142340
- [Derived] Katheria A, Reister F, Essers J, Mendler M, Hummler H, Subramaniam A, Carlo W, Tita A, Truong G, Davis-Nelson S, Schmolzer G, Chari R, Kaempf J, Tomlinson M, Yanowitz T, Beck S, Simhan H, Dempsey E, O'Donoghue K, Bhat S, Hoffman M, Faksh A, Arnell K, Rich W, Finer N, Vaucher Y, Khanna P, Meyers M, Varner M, Allman P, Szychowski J, Cutter G. Association of Umbilical Cord Milking vs Delayed Umbilical Cord Clamping With Death or Severe Intraventricular Hemorrhage Among Preterm Infants. JAMA. 2019 Nov 19;322(19):1877-1886. doi: 10.1001/jama.2019.16004. PMID 31742630
- See also: Website for trial — http://www.premod2.org
- See also: NIRS Sub-study PREMOD2 — https://clinicaltrials.gov/show/NCT03145142
- See also: Followup Study-PREMOD2 — http://clinicaltrials.gov/show/nct03476980